CLINICAL TRIAL: NCT06358209
Title: Safety and Efficacy of Ventricular Irrigation for Ventriculitis: a Randomized Controlled Trial
Brief Title: Safety and Efficacy of Ventricular Irrigation for Ventriculitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Southern Medical University, China (Other); First Affiliated Hospital of Zhejiang University (Other); 904th Hospital of the Joint Logistics Support Force of the PLA (Other); Shenzhen Second People's Hospital (Other); Shanghai East Hospital (Other); Xuanwu Hospital, Beijing (Other); South Taihu Hospital Affiliated to Huzhou College (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Yangzhou University (Other); The First Affiliated Hospital of Soochow University (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); West China Hospital (Other); The Second Affiliated Hospital of Air Force Medical University (Unknown); Qilu Hospital of Shandong University (Other); The Fourth Affiliated Hospital of China Medical University (Other); Ganzhou People's Hospital (Unknown); Xiangya Hospital of Central South University (Other); Tongji Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Henan Provincial People's Hospital (Other); The Second People's Hospital of Anhui Province (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); First Affiliated Hospital of Fujian Medical University (Other); Shanghai Donglei Brain Hospital (Unknown); The Affiliated People's Hospital of Ningbo University (Other Government); Inner Mongolia People's Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Affiliated Hospital of Nantong University (Other); The First Affiliated Hospital of Wannan Medical College（Yijishan Hospital of Wannan Medical College） (Unknown); The Second Affiliated Hospital of Naval Medical University (Shanghai Changzheng Hospital) (Unknown); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY2024-045-B
Record Dates: First submitted 2024-03-31; First posted 2024-04-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Infections
Keywords: Ventriculitis; Ventricular irrigation
MeSH Terms: conditions — Central Nervous System Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Conventional treatments for ventriculitis, including: external ventricular drainage or lumbar cistern drainage for continuous drainage, systemic and intrathecal antibiotics along with other supportive care. The treatment plan, including the type, dosage, and duration of antibiotics, follows guidelines "2017 Infectious Diseases Society of America's Clinical Practice Guidelines for Healthcare-Associated Ventriculitis and Meningitis" and "Chinese Expert Consensus on Diagnosis and Treatment of Central Nervous System Infections in Neurosurgery (2021 Edition)".
- Ventricular irrigation group (Experimental): Intervention group employs catheter ventricular irrigation with various forms. Lavage is performed with each time at least 200ml of normal saline, and irrigation treatment over 7 days. Additional treatments, including the administration of antibiotics, are consistent with those in the control group.
  Interventions: Procedure: Ventricular irrigation

INTERVENTIONS:
Procedure: Ventricular irrigation — Catheter ventricular irrigation can be employed by various forms. Lavage is performed with with each time at least 200ml of saline. Aside from lavage sessions, the lavage is paused, but continuous CSF drainage remains open.
  Arms: Ventricular irrigation group

SUMMARY:
Ventriculitis is a severe infectious disease of the central nervous system with diverse etiologies. Currently, the treatment for ventriculitis is challenging, with poor prognosis. The mortality rate of ventriculitis is generally reported to be higher than 30%, with the highest reaching over 75%. Even among survivors, over 60% suffer from a variety of neurological sequelae, including cognitive impairment, gait disturbances, paralysis, behavioral disorders, and epilepsy.

Currently, treatments for ventriculitis recommended by guidelines primarily focus on the selection and administration of antibiotics, while the effects of surgical interventions have not been fully elucidated. In recent years, several studies have explored the use of ventricular irrigation in ventriculitis, indicating that ventricular irrigation techniques may accelerate the control of ventricular infection, mitigate damage to the central nervous system caused by infections, improve the prognosis of ventriculitis, and reduce complications such as hydrocephalus. However, current studies are still relatively scarce, and mostly case reports and retrospective studies. High-quality evidence is still lacking for the application of ventricular irrigation in ventriculitis.

This multicenter randomized controlled trial aims to explore the safety and effectiveness of ventricular irrigation compared to conventional treatment for ventriculitis, analyze the effectiveness of ventricular irrigation across different pathogen subgroups, and investigate independent risk factors for different prognostic states in patients with ventriculitis.

DETAILED DESCRIPTION:
Ventriculitis is a severe infectious disease of the central nervous system with diverse etiologies. Ventriculitis is associated not only with community-acquired diseases but also, more importantly, with invasive clinical procedures, including craniotomy, external ventricular drainage (EVD), lumbar cistern drainage, V-P shunt, and deep brain stimulation, among others. Depending on the diagnostic criteria, the incidence of post-neurosurgery ventriculitis ranges from approximately 5% to 20%, with risk factors including age, prolonged placement of EVD, and intracranial hemorrhage. Besides, the pathogens leading to ventricular infection are also diverse, with the main pathogens including coagulase-negative Staphylococci, Staphylococcus aureus, Propionibacterium acnes, and Gram-negative bacilli.

The treatment for ventriculitis is challenging, with poor prognosis. Under currently widely adopted treatment strategies, the mortality rate of ventriculitis is generally reported to be higher than 30%, with the highest reaching over 75%. Even among survivors, over 60% suffer from a variety of neurological sequelae, including cognitive impairment, gait disturbances, paralysis, behavioral disorders, and epilepsy. This imposes significant burden on families and society. Therefore, how to further improve prognosis of ventriculitis, and reduce the mortality and disability rates, remains to be addressed.

Currently, treatments for ventriculitis recommended by guidelines primarily focus on the selection and administration of antibiotics, while the effects of surgical interventions have not been fully elucidated. As an infectious disease, surgical procedures such as irrigation and drainage have the potential to play a role in reducing infection and improving prognosis for ventriculitis.

In recent years, several studies have explored the use of ventricular irrigation in ventriculitis, indicating that ventricular irrigation techniques (including endoscopic ventricular irrigation and dual catheter irrigation techniques) via replacing saline and draining purulent cerebrospinal fluid (CSF), may accelerate the control of ventricular infection, mitigate damage to the central nervous system caused by infections, improve the prognosis of ventriculitis, and reduce complications such as hydrocephalus. However, current studies are still relatively scarce, and mostly case reports and retrospective studies. A prospective controlled study that included 33 patients with ventriculitis divided participants into groups receiving ventricular irrigation treatment and conventional treatment. The study results showed that compared to conventional treatment, ventricular irrigation resulted in higher mRS prognosis scores, shorter hospital stays, and the study also showed a trend towards reduced mortality in irrigation group. However, this study was limited by a small sample size, limited study endpoints and not strictly randomized. Currently, high-quality evidence is still lacking for the application of ventricular irrigation in ventriculitis.

Based on these considerations, this multicenter randomized controlled trial aims to explore the safety and effectiveness of ventricular irrigation compared to conventional treatment for ventriculitis, analyze the effectiveness of ventricular irrigation across different pathogen subgroups, and investigate independent risk factors for different prognostic states in patients with ventriculitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old;
* CSF is purulent (it appears cloudy or yellow) and white blood cell count over 1000×10^6/L.
* Fever (>38.0°C)
* Meet at least one of the following: 1. Patient has organism(s) identified from CSF by a culture or non-culture based microbiologic testing method; 2. Cranial CT or MRI indicating intraventricular floccule or pus.
* With consent form

Exclusion Criteria:

* With GCS score of 3
* With unstable vital signs such as no spontaneous breathing and blood pressure maintenance drugs
* With severe propensity for bleeding (Such as coagulation dysfunction, active bleeding, etc.), and unable to tolerate the surgical procedures or operations related to ventricular irrigation treatment.
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 4 weeks after enrollment
  Clinical cure rate at 4 weeks after enrollment and randomization

SECONDARY OUTCOMES:
GOSE | up 6 months after enrollment and randomization
  Extended Glasgow Outcome Scale at discharge and within 6 months after diagnosis of ventriculitis
CSF test results | At 8th day after enrollment, and within 1 week before discharge
  Results of CSF test at 8th day after enrollment, and within 1 week before discharge, including CSF glucose, CSF protein, CSF WBC count and organism(s) identification by a culture or non-culture based microbiologic testing method
Cranial CT or MRI indicating | At 8th day after enrollment, and within 1 week before discharge
  Cranial CT or MRI indicating at 8th day after enrollment, and within 1 week before discharge
Length of ICU stay and hospital stay | up to 6 months after enrollment and randomization
  Length of ICU stay and hospital stay
Complications | up to 6 months after enrollment and randomization
  Blood from puncture canal and intracranial during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jiyao Jiang, Dr, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Junfeng Feng, Dr, Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Qinghua Wang, Dr, Study Director — Southern Medical University, China; Xiaofeng Yang, Dr, Study Director — First Affiliated Hospital of Zhejiang University; Yuhai Wang, Dr, Study Director — 904th Hospital of the Joint Logistics Support Force of the PLA; Xianjian Huang, Dr, Study Director — Shenzhen Second People's Hospital; Xuefei Shao, Dr, Study Director — First Affiliated Hospital of Wannan Medical College; Lijun Hou, Dr, Study Director — The Second Affiliated Hospital of Naval Medical University; Chunlong Zhong, Dr, Study Director — Shanghai East Hospital; Liang Gao, Dr, Study Director — Shanghai Donglei Brain Hospital; Rongcai Jiang, Dr, Study Director — Xuanwu Hospital, Beijing; Liansheng Long, Dr, Study Director — South Taihu Hospital Affiliated to Huzhou College; Feng Gao, Dr, Study Director — he affiliated people's hospital of ningbo university; Chunhua Hang, Dr, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Jing Ji, Dr, Study Director — The First Affiliated Hospital with Nanjing Medical University; Xiaoou Sun, Dr, Study Director — The First Affiliated Hospital of Soochow University; Aijun Peng, Dr, Study Director — Yangzhou University; Jinlong Shi, Dr, Study Director — Affiliated Hospital of Nantong University; Binghui Qiu, Dr, Study Director — Nanfang Hospital, Southern Medical University; Dan Jin, Dr, Study Director — Zhongshan Hospital Of Traditional Chinese Medicine; Yongxin Wang, Dr, Study Director — First Affiliated Hospital of Xinjiang Medical University; Chaohua Yang, Dr, Study Director — West China Hospital; Qibing Huang, Dr, Study Director — Qilu Hospital of Shandong University; Yan Qu, Dr, Study Director — The Second Affiliated Hospital of Air Force Medical University; Yan Zhang, Dr, Study Director — Second Affiliated Hospital of Nanchang University; Qiuhua Jiang, Dr, Study Director — Ganzhou People's Hospital; Yijun Bao, Dr, Study Director — The Fourth Affiliated Hospital of China Medical University; Hongsheng Liang, Dr, Study Director — First Affiliated Hospital of Harbin Medical University; Wenhua Fang, Dr, Study Director — First Affiliated Hospital of Fujian Medical University; Guang Feng, Dr, Study Director — Henan Provincial People's Hospital; Kai Shu, Dr, Study Director — Tongji Hospital; Jinfang Liu, Dr, Study Director — Xiangya Hospital of Central South University; Weiping Zhao, Dr, Study Director — Inner Mongolia People's Hospital; Yongming Zhang, Dr, Study Director — The Second People's Hospital of Anhui Province; Xiangpin Wei, Dr, Study Director — The First Affiliated Hospital of University of Science and Technology of China; Xianzhen Chen, Dr, Study Director — Shanghai 10th People's Hospital
Locations (35):
- China (35):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - The Second People's Hospital of Anhui Province, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - 904 Hospital of the People's Liberation Army Joint Logistic Support Force, Wuxi, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Donglei Brain Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Inner Mongolia People's Hospital, Hohhot, The Nei Monggol Autonomous Region
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - South taihu hospital affiliated to huzhou college, Huzhou, Zhejiang
  - The affiliated people's hospital of ningbo university, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Researchers who submit a methodologically sound study proposal that is approved by the management committee can have access to the study protocol, individual participant data and data dictionary. A Data Access Agreement is required, and all access must comply with regulatory restrictions imposed on the original study.
Supporting Information: Study Protocol
Time Frame: After Publication
Access Criteria: Researchers who submit a methodologically sound study proposal that is approved by the management committee can have access to the study protocol, individual participant data and data dictionary.

REFERENCES:
- [Background] Tunkel AR, Hasbun R, Bhimraj A, Byers K, Kaplan SL, Scheld WM, van de Beek D, Bleck TP, Garton HJL, Zunt JR. 2017 Infectious Diseases Society of America's Clinical Practice Guidelines for Healthcare-Associated Ventriculitis and Meningitis. Clin Infect Dis. 2017 Mar 15;64(6):e34-e65. doi: 10.1093/cid/ciw861. PMID 28203777
- [Background] Al Menabbawy A, El Refaee E, Soliman MAR, Elborady MA, Katri MA, Fleck S, Schroeder HWS, Zohdi A. Outcome improvement in cerebral ventriculitis after ventricular irrigation: a prospective controlled study. J Neurosurg Pediatr. 2020 Sep 4;26(6):682-690. doi: 10.3171/2020.5.PEDS2063. Print 2020 Dec 1. PMID 32886918
- [Background] Hasbun R. Healthcare-associated ventriculitis: current and emerging diagnostic and treatment strategies. Expert Rev Anti Infect Ther. 2021 Aug;19(8):993-999. doi: 10.1080/14787210.2021.1866544. Epub 2020 Dec 24. PMID 33334204
- [Background] Humphreys H, Jenks PJ. Surveillance and management of ventriculitis following neurosurgery. J Hosp Infect. 2015 Apr;89(4):281-6. doi: 10.1016/j.jhin.2014.12.019. Epub 2015 Jan 29. PMID 25687249
- [Background] Rogers T, Sok K, Erickson T, Aguilera E, Wootton SH, Murray KO, Hasbun R. Impact of Antibiotic Therapy in the Microbiological Yield of Healthcare-Associated Ventriculitis and Meningitis. Open Forum Infect Dis. 2019 Feb 6;6(3):ofz050. doi: 10.1093/ofid/ofz050. eCollection 2019 Mar. PMID 30899767
- [Background] Karvouniaris M, Brotis A, Tsiakos K, Palli E, Koulenti D. Current Perspectives on the Diagnosis and Management of Healthcare-Associated Ventriculitis and Meningitis. Infect Drug Resist. 2022 Feb 28;15:697-721. doi: 10.2147/IDR.S326456. eCollection 2022. PMID 35250284
- [Background] Karvouniaris M, Brotis AG, Tsiamalou P, Fountas KN. The Role of Intraventricular Antibiotics in the Treatment of Nosocomial Ventriculitis/Meningitis from Gram-Negative Pathogens: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Dec;120:e637-e650. doi: 10.1016/j.wneu.2018.08.138. Epub 2018 Aug 29. PMID 30172065
- [Background] Luque-Paz D, Revest M, Eugene F, Boukthir S, Dejoies L, Tattevin P, Le Reste PJ. Ventriculitis: A Severe Complication of Central Nervous System Infections. Open Forum Infect Dis. 2021 Apr 29;8(6):ofab216. doi: 10.1093/ofid/ofab216. eCollection 2021 Jun. PMID 34095339
- [Background] Chan AK, Birk HS, Yue JK, Winkler EA, McDermott MW. Bilateral External Ventricular Drain Placement and Intraventricular Irrigation Combined with Concomitant Serial Prone Patient Positioning: A Novel Treatment for Gravity-Dependent Layering in Bacterial Ventriculitis. Cureus. 2017 Apr 18;9(4):e1175. doi: 10.7759/cureus.1175. PMID 28533993
- [Background] Terada Y, Mineharu Y, Arakawa Y, Funaki T, Tanji M, Miyamoto S. Effectiveness of neuroendoscopic ventricular irrigation for ventriculitis. Clin Neurol Neurosurg. 2016 Jul;146:147-51. doi: 10.1016/j.clineuro.2016.05.010. Epub 2016 May 9. PMID 27219537
- [Background] Gaderer C, Schaumann A, Schulz M, Thomale UW. Neuroendoscopic lavage for the treatment of CSF infection with hydrocephalus in children. Childs Nerv Syst. 2018 Oct;34(10):1893-1903. doi: 10.1007/s00381-018-3894-7. Epub 2018 Jul 11. PMID 29995267
- [Background] Qin G, Liang Y, Xu K, Xu P, Ye J, Tang X, Lan S. Neuroendoscopic lavage for ventriculitis: Case report and literature review. Neurochirurgie. 2020 Apr;66(2):127-132. doi: 10.1016/j.neuchi.2019.12.005. Epub 2020 Feb 19. PMID 32087178
- [Background] Stati G, Migliorino E, Moneti M, Castioni CA, Scibilia A, Palandri G, Virgili G, Aspide R. Treatment of cerebral ventriculitis with a new self-irrigating catheter system: narrative review and case series. J Anesth Analg Crit Care. 2023 Nov 8;3(1):46. doi: 10.1186/s44158-023-00131-5. PMID 37941074
- [Background] de Sousa Carvalho Dezena JE, Gerbelli CLB, Braga TKK, Ballestero MFM. How I do it: brainwashing for purulent ventriculitis. Acta Neurochir (Wien). 2023 Nov;165(11):3267-3269. doi: 10.1007/s00701-023-05607-5. Epub 2023 May 20. PMID 37209145
- [Background] Tomita Y, Shimazu Y, Kawakami M, Matsumoto H, Fujii K, Kameda M, Yasuhara T, Suruga Y, Ota T, Kimata Y, Kurozumi K, Date I. Pyogenic Ventriculitis After Anterior Skull Base Surgery Treated With Endoscopic Ventricular Irrigation And Reconstruction Using a Vascularized Flap. Acta Med Okayama. 2021 Apr;75(2):243-248. doi: 10.18926/AMO/61908. PMID 33953433
- [Background] Ochoa A, Arganaraz R, Mantese B. Neuroendoscopic lavage for the treatment of pyogenic ventriculitis in children: personal series and review of the literature. Childs Nerv Syst. 2022 Mar;38(3):597-604. doi: 10.1007/s00381-021-05413-3. Epub 2021 Nov 13. PMID 34775525